CLINICAL TRIAL: NCT05286112
Title: A Pilot Study on Mindfulness for Pain and Mental Health Outcomes
Brief Title: Mindfulness for Pain and Suicide
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Canandaigua VA Medical Center (U.S. Federal Agency)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1600604
Record Dates: First submitted 2022-01-28; First posted 2022-03-18 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Chronic Pain; Suicidal Ideation; Suicide, Attempted; Opioid Use
MeSH Terms: conditions — Chronic Pain; Suicidal Ideation; Suicide, Attempted | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Cognitive Therapy (MBCT) (Experimental): MBCT delivered over the course of 10, ~60 minute sessions
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy (MBCT)
- Health Education (Active Comparator): Health education sessions delivered over the course of 10, ~60 minute sessions
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy (MBCT) — 10 sessions focused on increasing mindfulness awareness to address thoughts, emotions, and behaviors that maintain functional impairment and risk of suicide.
  Arms: Mindfulness-Based Cognitive Therapy (MBCT)
Behavioral: Health Education — Health education provides information on the importance and benefits of and guidelines for living a healthy lifestyle.
  Arms: Health Education

SUMMARY:
The proposed study will assess the feasibility and acceptability of a mindfulness-based intervention to reduce functional impairment from chronic pain and risk of suicide.

DETAILED DESCRIPTION:
The investigators are seeking to develop a combined intervention, MBCT-S/P, to focus on both improving functioning and mitigating suicide risk in veterans with chronic pain. The investigators plan to test the new manual's feasibility and acceptability in a sample of veterans experiencing chronic pain and suicidal ideation. Participants will be randomized to either the MBCT-S/P condition (n=38) or the Education control condition (n=38) to assess additional aspects of study feasibility. The investigators also plan to assess a variety of clinical outcomes including suicidal ideation, pain interference in activities, and opioid use. Participants will complete questionnaires pre-treatment, and 1-, 3-, and 6-months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking veterans
* Ages 18 years and older
* Understand informed consent
* Report pain that occurs on at least half the days for six months or more
* Score at least a 4 on each item of the three items on a brief pain intensity and interference measure
* To meet the minimum threshold for suicide risk, veterans must meet at least one of the following: (1) endorse at least a 1 ("several days") on item 9 ("thoughts of you would be better off dead, or thoughts of hurting yourself in some way" in the past 2 weeks) of the Patient Health Questionnaire-9 (PHQ-9), (2) endorse at least "death ideation" in the last 3 months as measured by the Columbia Suicide Severity Rating Scale, or (3) report a suicide attempt in the last 6 months.

Exclusion Criteria:

* An active severe substance use disorder (SUD)
* Documented schizophrenia, active psychosis, or mania
* Upcoming surgeries
* Uncontrolled medical conditions
* Intent to carry out a plan for suicide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Treatment acceptability | 1-month post-treatment
  The Abbreviated Acceptability Rating Profile assesses the extent to which participants agree with 8 statements about the intervention. Scores range from 1 to 6 with higher scores indicating higher acceptability.
Suicide risk | baseline to 6 months post-treatment follow-up
  Suicide risk will be assessed using the Columbia Suicide Severity Rating Scale, which assesses presence and severity of suicidal ideation and behaviors in one's lifetime, over a specified period, and since the last visit. Presence of suicidal thoughts and behaviors are scored as either present (0) or absent (1) and severity is indicated as the most severe suicidal thought or behavior endorsed (from 0-none to 5-suicide attempt). Higher scores indicate more severe suicidal ideation and behaviors.
Depression | baseline to 6 months post-treatment follow-up
  The Patient Health Questionnaire-9, a 9-item measure assessing frequency of depression symptoms in the last week. Rating scale is from 0 to 3 with higher scores indicating more frequent depression symptoms.
Interpersonal Needs | baseline to 6 months post-treatment follow-up
  The Interpersonal Needs Questionnaire is a 12-item questionnaire measuring level of belonging and feeling like a burden to others. Items are rating on a scale ranging from 1 to 7 with higher scores indicate greater interpersonal conflict.
Pain Interference and intensity | baseline to 6 months post-treatment follow-up
  Pain interference and intensity will be measured using the Brief Pain Inventory. Four items assessing current, average, worst, and least pain experienced. Pain interference is assessed over 7 items across various life domains. Items are rated from 0 to 10 with higher scores indicating more severe pain intensity and greater interference in activities due to pain.

SECONDARY OUTCOMES:
Health-related Quality of Life | baseline to 6 months post-treatment follow-up
  The Veterans Rand (VR)-12 is a 12-item measure assessing health-related quality of life across physical (PCS) and mental health (MCS) components. PCS and MCS scores are derived using an algorithm that is referenced to a metric centered at 50.0. VR-12 scores are standardized using a T-score metric with a mean of 50 and a standard deviation of 10 with higher scores indicating better health-related quality of life.
Mindfulness | baseline to 6 months post-treatment follow-up
  The Five Facet Mindfulness Questionnaire (FFMQ) consists of 39 items that assess five elements of mindfulness: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. The rating scale ranges from 1 to 5 with higher scores indicated higher mindfulness.
Pain acceptance | baseline to 6 months post-treatment follow-up
  The Chronic Pain Acceptance Questionnaire (CPAQ) is a 20-item measure that assesses two components of pain acceptance: pursuit of life activities regardless of pain and recognition that avoidance is not useful in adapting to chronic pain. The rating scale ranges from 0 to 6 with higher scores indicating greater pain acceptance.
Pain catastrophizing | baseline to 6 months post-treatment follow-up
  The Pain Catastrophizing Scale (PCS) is a 13-item measure, with each item rated on a 5-point rating scale (0 = "Not at all" to 4 = "All the time"). The measure is divided into three subscales: magnification, rumination, and helplessness. Higher scores indicate greater pain catastrophizing.
Pain-related self-efficacy | baseline to 6 months post-treatment follow-up
  The Pain Self-efficacy Questionnaire (PSEQ) assesses one's confidence in performing activities while in pain. The rating scale ranges from 0 to 6 with higher scores indicating greater self-efficacy.
Fear of pain | baseline to 6 months post-treatment follow-up
  The Tampa Scale of Kinesiophobia-11 (TSK) is an 11-item measure assessing pain-related fear of movement or injury. The rating scale ranges from 1 to 4 with high scores indicating greater fear of movement.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Veterans Affairs Center of Excellence for Suicide Prevention, Canandaigua, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant data is available upon request as part of scientific collaboration.